CLINICAL TRIAL: NCT06437535
Title: The Pathophysiological Role of Vaspin and Apoptosis in Pre-eclamptic Obese Women
Brief Title: Role of Vaspin in Pathophysiology of Pre-eclampsia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ali Ibrahim Sayed, principal investigator, Assiut University
Other Study IDs: vaspin and pre-eclampsia
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: will include 25 women with normal weight and normal blood pressure .
- Group2: :will include 25 obsese women with normal blood pressure.
- Group 3: : will include 25 obese women with confirmed diagnosis of severe preeclampsia .

SUMMARY:
* To investigate the possible role of vaspin and apoptosis in pre-eclamptic obese women .
* To compare the serum as well as placental level of vaspin in normotensive and severe pre-eclamptic obese women.
* To compare the serum as well as placental level of vaspin in normotensive normal body weight and severe pre-eclamptic obese women women .
* To compare placental apoptosis marker Bcl2 in normotensive and severe pre-eclamptic obese women .
* To compare placental apoptosis marker Bcl2 in normotensive normal body weight and severe pre-eclamptic obese women .
* Correlation between vaspin and apoptosis in pre-eclamptic obese women .
* Correlation between vaspin level and apoptosis marker with patient demographic data(Age -parity).

DETAILED DESCRIPTION:
• Pre-eclampsia(PE) is defined as new onset hypertension after 20 weeks gestation with evidence of maternal organ or uteroplacental dysfunction or proteinuria. The majority of maternal deaths related to PE can be avoided by providing timely and effective care and delivery to high-risk women. Thus, optimization of health care for women during pregnancy to prevent and treat PE . PE classified clinically to mild and severe sub types as Pregnant women with BP≥160/110 mmHg and proteinuria ≥3+ reading on dipstick are classified as having severe PE while pregnant women with systolic blood pressure of 140 -159 mmHg, diastolic blood pressure of 90-109 mmHg, and proteinuria ≥1+ reading on dipstick are classified as having mild PE.. Vaspin, a member of adipokines was first isolated from the visceral adipose tissue of the rat abdominal obesity model (OLETF). It belongs to the serine protease inhibitors and acts through a protein G-coupled receptor - GRP78. Vaspin has also found in the liver, pancreas, cerebrospinal ﬂuid, hypothalamus, intestine, and lungs.it has pleiotropic functions that include regulating inﬂammatory response, insulin resistance and the development of obesity. Vaspin like other adipokines including leptin and adiponectin can aﬀect the female reproduction system like ovary. Vaspin expression was detected in another reproductive component, the placenta. In humans, vaspin was localized in cytotrophoblasts and syncytiotrophoblasts in ﬁrst-trimester placentas, but only in syncytiotrophoblasts in third-trimester placentas. Apoptosis plays a critical role in the homeostasis regulation of normal placental development. However, excessive placental apoptosis leads to placental dysfunction, which may consequence in pregnancy disorders such as preeclampsia. vaspin acts as an antiapoptotic agent in ovary by attenuating the tumor necrosis factor (TNF-α)-induced apoptosis by promoting autophagy also has been shown to inhibit macrophage apoptosisAnti apoptotic eﬀects of vaspin have also been described in human osteoblast cells by upregulation of the expression of BCL2 and downregulation of BAX through the Mitogen-activated kinase (MAP3/1)pathway and Protein kinase B(AKT) pathway.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women who will come to hospital for termination of pregnancy .
* Confirmed diagnosis of preeclampsia for study groups.
* Control group will include Normotensive pregnant women.
* Age group 18-35 years.
* gestional age at termination of pregnancy : group 1&2 : from 38 to 40 weeks group 3:terminatin of pregnancy regardless of gestional age

Exclusion Criteria:

* Pregnant women who do not consent to participate.
* Diabeteic patients .
* History of pre-gestional hypertension.
* History of chronic renal disease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women who will come for termination of pregnancy
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
vaspin level in serum and placenta | one year
  - measure level of vaspin in serum as well as its level in placenta in patients with pre-eclampsia and women with normal pregnancy
level of bcl2 expression in placenta | one year
  measure level of gene expression of apoptotic marker bcl2 by PCR in placenta in patients with preeclampsia and women with normal pregnancy
vaspin and bcl2 | one year
  correlation between level of vaspin and bcl2 gene expression in patients of preeclamsia and women with normal pregnancy

SECONDARY OUTCOMES:
vapin level and bcl2 level and patient demographic data | one year
  Correlation between vaspin level and bcl2 level with patient demographic data(Age -parity).

REFERENCES:
- [Background] Bergman L, Torres-Vergara P, Penny J, Wikstrom J, Nelander M, Leon J, Tolcher M, Roberts JM, Wikstrom AK, Escudero C. Investigating Maternal Brain Alterations in Preeclampsia: the Need for a Multidisciplinary Effort. Curr Hypertens Rep. 2019 Aug 2;21(9):72. doi: 10.1007/s11906-019-0977-0. PMID 31375930
- [Background] Fondjo LA, Sarpong D, Owiredu WKBA, Opoku S, Adu-Bonsaffoh K, Teviu E. Effect of magnesium sulfate treatment on mediators of endothelial dysfunction and electrolytes in mild and severe preeclampsia: A case-control study. Health Sci Rep. 2023 Apr 26;6(5):e1232. doi: 10.1002/hsr2.1232. eCollection 2023 May. PMID 37123551
- [Background] Kurowska P, Mlyczynska E, Dawid M, Jurek M, Klimczyk D, Dupont J, Rak A. Review: Vaspin (SERPINA12) Expression and Function in Endocrine Cells. Cells. 2021 Jul 6;10(7):1710. doi: 10.3390/cells10071710. PMID 34359881
- [Background] Kurowska P, Mlyczynska E, Dawid M, Opydo-Chanek M, Dupont J, Rak A. In Vitro Effects of Vaspin on Porcine Granulosa Cell Proliferation, Cell Cycle Progression, and Apoptosis by Activation of GRP78 Receptor and Several Kinase Signaling Pathways Including MAP3/1, AKT, and STAT3. Int J Mol Sci. 2019 Nov 19;20(22):5816. doi: 10.3390/ijms20225816. PMID 31752432